CLINICAL TRIAL: NCT07049562
Title: Study on the Mass Balance of [14C]HRS-8427 for Injection in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8427-104
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Healthy Cninese Adult Male

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A: [14C] HRS-8427 (Experimental)
  Interventions: Drug: HRS-8427

INTERVENTIONS:
Drug: HRS-8427 — [14C] HRS-8427 for injection

SUMMARY:
To evaluate the absorption, metabolism and excretion after a single intravenous infusion of [14C]HRS-8427 in healthy Chinese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male ages 18~45 years, inclusive;
2. The body weight should be no less than 50 kg, and the body mass index (BMI) should be within the range of 19.0 kg/m2 to 26.0 kg/m2, inclusive;
3. Subjects without sperm donation or fertility plan, and agree to adopt highly medically effective contraceptive measurements during the trial and within 3 months after the last dose;
4. Participants voluntarily sign the informed consent form before the trial, can communicate well with the researcher, have a full understanding of the trial content, process and possible adverse reactions, and can complete the trial in accordance with the protocol.

Exclusion Criteria:

1. A history of allergies to food, drugs allergic constitution;
2. History or presence of seriousmediacl diseases judged by the investigator as not suitable for the study;
3. Perianal diseases with regular or ongoing bloody stools, irritable bowel syndrome, and inflammatory bowel disease;
4. Habitual constipation or diarrhea;
5. Those who have undergone major surgical operations within the three months prior to screening; Or those who have undergone surgery that may affect the in vivo process or safety evaluation of the studied drug; Or those who plan to undergo surgical operations during the research period;
6. With abnormal and clinically significant comprehensive physical examinations, vital signs, or laboratory examinations
7. Abnormal 12-lead electrocardiogram and determined by the researcher as unsuitable to participate in this study
8. Tested positive for HIV antibodies, hepatitis B surface antigen, hepatitis C, or Treponema pallidum antibodies;
9. Those who have used other clinical trial drugs within 3 months before the trial or plan to participate in other clinical trials during this study period;
10. Those have experienced blood loss or donated up to 300 mL of blood, or have received blood transfusion or used blood products, or plan to donate blood during the trial or within 1 month after the end of the trial;
11. Abuse of alcohol or drugs
12. Heavy smokers or caffeine addicts.
13. Those engaged in long-term exposure to radioactive conditions; Or those who have had significant radioactive exposure within one year before the test or have participated in radiopharmaceutical tests within one year;
14. Those who cannot accept a uniform diet or have special dietary requirements;
15. Participants who may be unable to complete this study for other reasons or who the researcher deems should not be included.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
The total radioactive recovery rate and cumulative total radioactive recovery rate at each time interval in excreta (urine and feces) | 0~120hours
The percentage (%AUC) of the potent drug and its metabolites in plasma, urine and feces to the administered dose | 0~120hours
Tmax | 0~48hours
Cmax | 0~48hours
t1/2 | 0~48hours
MRT | 0~48hours
AUC | 0~48hours

SECONDARY OUTCOMES:
Tmax | 0~48hours
Cmax | 0~48hours
MRT | 0~48hours
AUC | 0~48hours
t1/2 | 0~48hours
Adverse events | 0~120hours

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided